CLINICAL TRIAL: NCT06530485
Title: Enhancing Immunity and Nutrition in Severely Malnourished Children Following Hospital Discharge: a Two Arm Open-label Randomized Controlled Trial of Microbiota-Directed Food vs. Zinc With Micronutrient Powder and Khichuri
Brief Title: Post Discharge Trial to Enhance Immunity in Severely Malnourished Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR-24010
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-06

CONDITIONS: Child Malnutrition
Keywords: Immunity; Malnutrition; Microbiota-directed food (MDF); Zinc; NK cells; Gut microbiota
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — milk-derived factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiota-directed food (Experimental): Children randomized to this group will receive Microbiota-directed food (MDF) daily for 12 weeks. MDF can modulate the gut microbiota and enhance host immunity, growth, and development in malnourished children.
  Interventions: Dietary Supplement: Microbiota-directed food
- Khichuri (Active Comparator): Children randomized to this group will receive zinc with Micronutrient powder (MNP) and Khichuri daily for 12 weeks.
  Interventions: Dietary Supplement: Khichuri

INTERVENTIONS:
Dietary Supplement: Microbiota-directed food — MDF can modulate the gut microbiota and enhance host immunity, growth, and development in malnourished children. Each sachet of MDF (100 gm) provides approximately 500 kcal.
  Other Names: MDF
  Arms: Microbiota-directed food
Dietary Supplement: Khichuri — Khichuri is a home-based nutritious food with high energy and protein. This arm also contains zinc (10 gm/day), micronutrient powder, and an egg daily.
  Other Names: Locally available food
  Arms: Khichuri

SUMMARY:
The goal of this study is to evaluate the efficacy of microbiota-directed food in comparison to zinc with micronutrient powder and Khichuri on changes in circulating immune cells (monocytes, T cells, B cells, and NK cells) in malnourished children after recovery from acute infection.

The study aims to answer the research question:

Does microbiota-directed food (MDF) compared to zinc with micronutrient powder (MNP) and Khichuri therapy enhance immunity in children with severe acute malnutrition? The researcher will compare the effectiveness of microbiota-directed food (MDF) versus zinc with micronutrient powder (MNP) and Khichuri therapy to see if MDF enhances immunity in severely malnourished children.

Severely malnourished children will:

* Receive microbiota-directed food (MDF) or zinc with micronutrient powder (MNP) and Khichuri every day for 12 weeks.
* Phenotyping of circulating immune cells (NK cells, T cells, B cells) will be conducted using flow cytometry and fluorescence-activated cell sorting techniques.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 36 months, and
* Severe acute malnutrition as evident by weight-for-length z-score (WLZ) < -3 and or mid-upper arm circumference (MUAC) < 11.5 cm, and or edema of both feet, and
* Completed the acute phase management for SAM and stayed at NRU for 7±4 days, with no medical complications, e.g. lethargic/unconscious, convulsions, unable to drink, persistent vomiting, respiratory distress.
* Residing within the Dhaka district.
* Parents/guardians provided written informed consent.

Exclusion Criteria:

* WLZ ≥ -3 or MUAC ≥11.5 cm.
* Presence of lethargy/unconsciousness, convulsions, unable to drink, persistent vomiting, respiratory distress.
* Participants who receive multiple courses of antibiotic (>2 courses during acute phase) treatment for a prolonged period (>14 days).
* Persistent diarrhea (≥14 days).
* Chronic illness or disability affecting food intake, e.g. TB, HIV, congenital defects, cerebral palsy
* Treated for SAM in the previous 3 months.
* Known case of soy, peanut, or milk protein allergy.
* Any sibling of the enrolled child.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NK cells | 12 weeks
  Differences in the proportion and activity of circulating NK cells between the groups 12 weeks after the intervention, measured by flow cytometry/fluorescence-assisted cell sorter (FACS).

SECONDARY OUTCOMES:
Circulating immune cells | 12 weeks
  Differences in the proportion of circulating immune cells (NK cells, T cells, B cells) before and after the interventions
Cytokines and chemokines | 12 weeks
  Differences in the levels of pro-inflammatory and anti-inflammatory cytokines and chemokines in circulation, which can provide insights into the functional status of immune cells
Micro biocidal capacity | 12 weeks
  Differences in the micro biocidal capacity (oxidative burst) of neutrophils and monocytes.
Rate of weight gain | 12 weeks
  Rate of weight gain between the intervention groups over the 12-weeek intervention period.
Diarrhea and pneumonia | 12 weeks
  Incidence of acute diarrhea and pneumonia during the study period.
Gut microbiota | 12 weeks
  Composition and evolution of gut microbiota over the 12-weeek intervention period.
Case fatality rate | 12 weeks
  Case fatality rate within 12 weeks post discharge.
Anthropometric recovery | 12 weeks
  Anthropometric recovery from SAM: anthropometric recovery will be defined as reaching a WLZ of >-2 (for those admitted with WLZ <-2) and or MUAC >12.5 (for those admitted with MUAC <12.5 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Farzana Afroze, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

IPD SHARING:
Plan to Share IPD: No